CLINICAL TRIAL: NCT02883972
Title: Can Uptake of Childhood Influenza Immunisation Through Schools be Increased Through Behavioural-insight Informed Changes to the Invitation Process?
Brief Title: Childhood Influenza Immunisation Invitation Trial in Schools
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethical approval was withdrawn by the National Research Ethics Service as they were unable to make contact with the research team despite trying many times.
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2016_FluInvSch
Record Dates: First submitted 2016-07-22; First posted 2016-08-30 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2016-07

CONDITIONS: Influenza, Human
Keywords: Immunization; Behavioural insights; Children
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention letter and reminder (Experimental): Behavioural insights informed invitation letter and SMS/email reminder message
  Interventions: Other: Intervention letter; Other: Reminder
- Intervention letter (Experimental): Behavioural insights informed invitation letter only
  Interventions: Other: Intervention letter
- Control letter and reminder (Experimental): Control invitation letter and SMS/email reminder message
  Interventions: Other: Control letter; Other: Reminder
- Control letter (Active Comparator): Control invitation letter only
  Interventions: Other: Control letter

INTERVENTIONS:
Other: Intervention letter — Behavioural-insight informed letter template
  Arms: Intervention letter; Intervention letter and reminder
Other: Control letter — Invitation letter used by local area last year (updated as required)
  Arms: Control letter; Control letter and reminder
Other: Reminder — Behavioural-insight informed SMS/email reminder message to return consent form
  Arms: Control letter and reminder; Intervention letter and reminder

SUMMARY:
This study will investigate whether influenza vaccine uptake by school-age children (in school-based clinics) can be increased by making behavioural-insight informed changes to the invitation process which encourage parents to return consent forms.

DETAILED DESCRIPTION:
Previous research has shown that small changes to the invitation phrasing and/or process informed by understanding and insights into behaviour can be used to increase a desired behaviour (e.g. uptake of health checks, reducing primary care antibiotic prescribing).

This trial will determine whether a behaviour-insight informed invitation letter and/or reminder Short Message Service (SMS)/email message can increase return of consent forms and thereby increase uptake of childhood flu vaccine in schools.

The trial will take place within the existing national childhood immunisation programme in participating areas in England. Randomisation will be at the school-level (stratified by local authority). All eligible children within a school will therefore be in the same arm of the trial and be subject to the same invitation process. Outcome data will be routinely collected, school-level influenza vaccine uptake data. Data will also be collected on the implementation of email/SMS reminders in all schools.

The analysis will investigate the main effects of the interventions and their interactions, take into account provider, local authority and school effects and explore the impact of other factors such as deprivation indicators.

An analysis of letters used by providers of childhood influenza immunisation in schools not involved in the trial will also be conducted. All providers will be asked to submit a copy of their invitation letter for the 2016/17 programme and these will be analysed using the Theoretical Domains Framework.

ELIGIBILITY:
Inclusion Criteria:

* Attendance at a school where national childhood influenza immunisation programme is delivered by a provider participating in the trial
* Eligible for influenza immunisation

Exclusion Criteria:

* Ineligible for influenza immunisation

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Influenza immunisation uptake in school years 1-3 | 5 months
  Proportion of children in school years 1-3 who receive influenza immunisation as part of the national childhood immunisation programme

SECONDARY OUTCOMES:
Influenza immunisation uptake in school years 4-6 | 5 months
  Proportion of children in school years 4-6 who receive influenza immunisation
Influenza immunisation uptake in Reception school year | 5 months
  Proportion of children in Reception school year who receive influenza immunisation
Influenza immunisation uptake in each school year | 5 months
  Proportion of children in each school year who receive influenza immunisation
Influenza immunisation consent in school years 1-3 | 5 months
  Proportion of children in school years 1-3 for who consent is neither given nor withheld (i.e. non-responders)
Influenza immunisation consent in school years 4-6 | 5 months
  Proportion of children in school years 4-6 for who consent is neither given nor withheld (i.e. non-responders)
Influenza immunisation consent in Reception school year | 5 months
  Proportion of children in Reception school year for who consent is neither given nor withheld (i.e. non-responders)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Chadborn, BSc MSc PhD, Principal Investigator — Public Health England

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howell-Jones R, Gold N, Bowen S, Bunten A, Tan K, Saei A, Jones S, MacDonald P, Watson R, Bennett KF, Chadborn T. Can uptake of childhood influenza immunisation through schools and GP practices be increased through behaviourally-informed invitation letters and reminders: two pragmatic randomized controlled trials. BMC Public Health. 2023 Jan 20;23(1):143. doi: 10.1186/s12889-022-14439-4. PMID 36670376

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT02883972/Prot_SAP_000.pdf